CLINICAL TRIAL: NCT01307319
Title: Study of Two Doses of an Investigational Nasal Aerosol Placebo Nasal Aerosol in Children (Ages 6-11) With Seasonal Allergies
Brief Title: Study of an Investigational Nasal Aerosol or Placebo Nasal Aerosol in Children (Ages 6-11) With Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-AR-305
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Seasonal Allergic Rhinitis; SAR
Keywords: Allergies; Hayfever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — alpha-ketoisovalerate dehydrogenase phosphatase; Beclomethasone; apaflurane; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BDP HFA 80 mcg/day (Experimental): Participants/parents administer 40 mcg of beclomethasone dipropionate hydrofluoroalkane (BDP HFA) (one spray per nostril) once daily for 15 days.
  Interventions: Drug: BDP HFA
- BDP HFA 160 mcg/day (Experimental): Participants/parents administer 80 mcg of beclomethasone dipropionate hydrofluoroalkane (BDP HFA) (one spray per nostril) once daily for 15 days.
  Interventions: Drug: BDP HFA
- Placebo nasal aerosol once daily (Placebo Comparator): Participants/parents administer placebo (a spray with no medication in each nostril) once daily for 15 days.
  Interventions: Drug: Placebo nasal aerosol

INTERVENTIONS:
Drug: BDP HFA — BDP (beclomethasone dipropionate) HFA (hydrofluoroalkane) nasal aerosol administered as a single actuation in each nostril daily for the 15 day treatment period. Each actuation contains either 40 or 80 mcg for a total daily dose of either 80 or 160 mcg depending upon the assigned treatment arm.
  Other Names: BDP (beclomethasone dipropionate) HFA (hydrofluoroalkane) Nasal Aerosol; QNASL®
  Arms: BDP HFA 160 mcg/day; BDP HFA 80 mcg/day
Drug: Placebo nasal aerosol — Placebo formulated as a nasal aerosol spray and administered as a single actuation in each nostril daily for the 15 day treatment period.
  Arms: Placebo nasal aerosol once daily

SUMMARY:
The purpose of this study is to assess the safety and efficacy of an investigational nasal aerosol at two doses compared with placebo nasal aerosol in the treatment of seasonal allergic rhinitis in children (6-11 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 6 to 11 years of age, as of the Screening Visit (SV)
* A documented history of SAR to a relevant seasonal allergen (tree/grass pollen) for a minimum of two years immediately preceding the study Screening Visit (SV).
* A demonstrated sensitivity to at least one seasonal allergen (tree/grass pollen) known to induce SAR through a standard skin prick test.
* Other criteria apply

Exclusion Criteria:

* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma (e.g., nasal piercing) or surgery, atrophic rhinitis, or rhinitis medicamentosa (all within the last 60 days prior to the Screening Visit [SV])
* History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, chronic sinusitis or influenza,) within the 14 days preceding the Screening Visit (SV), or development of a respiratory infection during the Run-in Period.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drug (e.g., theophylline, leukotriene antagonists). History of intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists prior to the Screening Visit (SV) is acceptable
* Have any conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial
* Other criteria apply

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 715 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Teva Clinical Study Site, Oxford, Alabama
  - Teva Clinical Study Site, Bell, California
  - Teva Clinical Study Site, Costa Mesa, California
  - Teva Clinical Study Site, Mission Viejo, California
  - Teva Clinical Study Site, Orange, California
  - Teva Clinical Study Site, Paramount, California
  - Teva Clinical Study Site, San Diego, California
  - Teva Clinical Study Site, Stockton, California
  - Teva Clinical Study Site, Centennial, Colorado
  - Teva Clinical Study Site, Colorado Springs, Colorado
  - Teva Clinical Study Site, Gainesville, Georgia
  - Teva Clinical Study Site, Lawrenceville, Georgia
  - Teva Clinical Study Site, Savannah, Georgia
  - Teva Clinical Study Site, Stockbridge, Georgia
  - Teva Clinical Study Site, Indianapolis, Indiana
  - Teva Clinical Study Site, Bethesda, Maryland
  - Teva Clinical Study Site, Minneapolis, Minnesota
  - Teva Clinical Study Site, Plymouth, Minnesota
  - Teva Clinical Study Site, Columbia, Missouri
  - Teva Clinical Study Site, Rolla, Missouri
  - Teva Clinical Study Site, Warrensburg, Missouri
  - Teva Clinical Study Site, Bozeman, Montana
  - Teva Clinical Study Site, Brick, New Jersey
  - Teva Clinical Study Site, High Point, North Carolina
  - Teva Clinical Study Site, Oklahoma City, Oklahoma
  - Teva Clinical Study Site, Portland, Oregon
  - Teva Clinical Study Site, Blue Bell, Pennsylvania
  - Teva Clinical Study Site, Collegeville, Pennsylvania
  - Teva Clinical Study Site, Philadelphia, Pennsylvania
  - Teva Clinical Study Site, Pittsburgh, Pennsylvania
  - Teva Clinical Study Site, Charleston, South Carolina
  - Teva Clinical Study Site, Orangeburg, South Carolina
  - Teva Clinical Study Site, Austin, Texas
  - Teva Clinical Study Site, Dallas, Texas
  - Teva Clinical Study Site, El Paso, Texas
  - Teva Clinical Study Site, Fort Worth, Texas
  - Teva Clinical Study Site, Houston, Texas
  - Teva Clinical Study Site, Kerrville, Texas
  - Teva Clinical Study Site, New Braunfels, Texas
  - Teva Clinical Study Site, San Antonio, Texas
  - Teva Clinical Study Site, Waco, Texas
  - Teva Clinical Study Site, Burke, Virginia
  - Teva Clinical Study Site, Richmond, Virginia

REFERENCES:
- [Derived] Storms WW, Segall N, Mansfield LE, Amar NJ, Kelley L, Ding Y, Tantry SK. Efficacy and safety of beclomethasone dipropionate nasal aerosol in pediatric patients with seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2013 Nov;111(5):408-414.e1. doi: 10.1016/j.anai.2013.07.033. Epub 2013 Aug 28. PMID 24125150

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1026 subjects were screened and 906 were enrolled and participated in the Run-in Period. Of the 906 enrolled subjects, 715 were randomized to treatment.
Period: Overall Study
Arm/Group | BDP HFA 80 mcg/Day | BDP HFA 160 mcg/Day | Placebo Nasal Aerosol Once Daily
Started | 239 (Randomized) | 242 (Randomized) | 234 (Randomized)
Safety Population | 239 | 241 (One participant was randomized in error and did not receive study medication.) | 234
ITT Population | 238 (One participant provided no post-baseline assessment.) | 241 | 234
Completed | 235 | 234 | 227
Not Completed | 4 | 8 | 7
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Other | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety population: the safety population included all randomized participants who received at least one dose of randomized study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP HFA 80 mcg/Day | BDP HFA 160 mcg/Day | Placebo Nasal Aerosol Once Daily | Total
Number analyzed (Participants) | 239 | 241 | 234 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.73) | 9.1 (1.62) | 9.1 (1.65) | 9.0 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 116 | 111 | 332
  Male | 134 | 125 | 123 | 382
Race/Ethnicity, Customized [Number; unit: participants]
  White | 169 | 172 | 164 | 505
  Black or African American | 56 | 55 | 52 | 163
  Asian | 2 | 4 | 6 | 12
  Other | 12 | 10 | 12 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 40 | 53 | 45 | 138
  Not Hispanic or Latino | 199 | 188 | 189 | 576
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.0 (4.15) | 19.4 (4.52) | 19.1 (4.72) | 19.1 (4.46)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Instantaneous Total Nasal Symptom Score (iTNSS) During the Two Weeks of Treatment
Description: Instantaneous TNSS is an evaluation of symptom severity over the last 10 minutes prior to the recording of the score. Participants (with assistance from parents/guardians/caregivers, as needed) assessed and recorded four nasal symptoms (runny nose, nasal congestion, nasal itching, and sneezing) twice daily (AM and PM) using the following scale:
  * 0 = absent (no sign/symptom present)
  * 1 = mild (sign/symptom clearly present, but minimal awareness; easily tolerated)
  * 2 = moderate (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping) The total TNSS scale was 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms.
  Baseline was defined as the average AM and PM subject-reported iTNSS over the 4 days prior to randomization.
Time Frame: Baseline (Day -4 to Day 1 predose), Days 1 (postdose) to Day 15
Population: The intent to treat (ITT) population included all randomized participants who received at least one dose of randomized study medication and had at least one post-baseline assessment. Two enrolled participants were excluded. One was randomized in error and did not receive test medication. The other provided no post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 mcg/Day | BDP HFA 160 mcg/Day | Placebo Nasal Aerosol Once Daily
Number analyzed (Participants) | 238 | 241 | 234
units on a scale | -1.6 (0.13) | -1.7 (0.13) | -1.0 (0.13)
Statistical Analysis 1: Comparison: BDP HFA 80 mcg/Day vs Placebo Nasal Aerosol Once Daily; Test type: Superiority or Other; p < 0.001, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.63, 95% CI 2-sided [-1.0 to -0.3]
Statistical Analysis 2: Comparison: BDP HFA 160 mcg/Day vs Placebo Nasal Aerosol Once Daily; Test type: Superiority or Other; p < 0.001, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.73, 95% CI 2-sided [-1.1 to -0.4]

2. Primary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Reflective Total Nasal Symptom Score (rTNSS) During the Two Weeks of Treatment
Description: Reflective TNSS is an evaluation of symptom severity over the past 12 hours prior to the recording of the score. Participants (with assistance from parents/guardians/caregivers, as needed) assessed and recorded four nasal symptoms (runny nose, nasal congestion, nasal itching, and sneezing) twice daily (AM and PM) using the following scale:
  * 0 = absent (no sign/symptom present)
  * 1 = mild (sign/symptom clearly present, but minimal awareness; easily tolerated)
  * 2 = moderate (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping) The total TNSS scale was 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms.
  Baseline was defined as the average AM and PM subject-reported rTNSS over the 4 days prior to randomization.
Time Frame: Baseline (Day -4 to Day 1 predose), Days 1 (postdose) to Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 mcg/Day | BDP HFA 160 mcg/Day | Placebo Nasal Aerosol Once Daily
Number analyzed (Participants) | 238 | 241 | 234
units on a scale | -1.9 (0.14) | -2.0 (0.14) | -1.2 (0.14)
Statistical Analysis 1: Comparison: BDP HFA 80 mcg/Day vs Placebo Nasal Aerosol Once Daily; The power calculation assumed the standard deviation (SD) for the change from baseline over two weeks in the average of AM and PM reflective TNSS is assumed to be 2.0. Using this standard deviation, 235 subjects per arm provides 90% power to detect a difference of 0.60 in TNSS change from baseline between treatment groups with a two-sided alpha level of 0.05; Test type: Superiority or Other; p < 0.001, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.71, 95% CI 2-sided [-1.1 to -0.3]
Statistical Analysis 2: Comparison: BDP HFA 160 mcg/Day vs Placebo Nasal Aerosol Once Daily; Test type: Superiority or Other; p < 0.001, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.76, 95% CI 2-sided [-1.1 to -0.4]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 6
Arm/Group | BDP HFA 80 mcg/Day | BDP HFA 160 mcg/Day | Placebo Nasal Aerosol Once Daily
Serious Adverse Events (participants affected / at risk) | 0/239 | 0/241 | 0/234
Other Adverse Events (participants affected / at risk) | 0/239 | 0/241 | 0/234

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.